CLINICAL TRIAL: NCT00026377
Title: A Phase I Study Of SU5416 With Androgen Ablation And Radiation In Patients With Intermediate and Advanced Stage Prostate Cancer
Brief Title: SU5416 Plus Hormone Therapy and Radiation Therapy in Treating Patients With Prostate Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11193A; UCCRC-NCI-4390; NCI-4390
Record Dates: First submitted 2001-11-09; First posted 2004-02-06 (Estimated); Last update posted 2013-09-05 (Estimated); Status verified 2013-09

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; stage IIB prostate cancer; stage IIA prostate cancer; stage III prostate cancer; stage IV prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — bicalutamide; Flutamide; Goserelin; Leuprolide; Semaxinib; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SU5416 in combination with hormone and radiation therapy (Experimental): Subjects receive 5 months of hormone suppression therapy consisting of 1 month of Bicalutamide or Flutamide followed by 4 months of leuprolide or goserlin injections. After completion of at least 12 weeks of hormone therapy, subjects will receive 7 1/2 weeks of radiation therapy. SU5416 will be given by IV infusion starting 4 weeks before beginning radiation treatment and continuing until 4 weeks after completion of radiation. Multiple doses of SU5416 will be studied.
  Interventions: Drug: bicalutamide; Drug: flutamide; Drug: goserelin acetate; Drug: leuprolide acetate; Drug: SU5416; Radiation: radiation therapy

INTERVENTIONS:
Drug: bicalutamide — 50 mg daily for 1 month
Drug: flutamide — 250 mg 3 times daily for 1 month
Drug: goserelin acetate — 3.6 mg once a month for 4 months
Drug: leuprolide acetate — 7.5 mg once a month for 4 months
Drug: SU5416 — IV infusion at assigned dose
Radiation: radiation therapy — daily for 5 days each week

SUMMARY:
RATIONALE: SU5416 may stop the growth of cancer by stopping blood flow to the tumor. Androgens can stimulate the growth of prostate cancer cells. Hormone therapy using flutamide, bicalutamide, leuprolide, or goserelin may fight prostate cancer by reducing the production of androgens. Radiation therapy uses high-energy x-rays to damage tumor cells. Combining SU5416, hormone therapy, and radiation therapy may kill more tumor cells.

PURPOSE: Phase I trial to study the effectiveness of SU5416 plus hormone therapy and radiation therapy in treating patients who have prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the safety of SU5416 in combination with standard androgen ablation and radiotherapy in patients with intermediate or advanced-stage prostate cancer.

OUTLINE: This is a multicenter, dose-escalation study of SU5416. Patients receive oral bicalutamide once daily or oral flutamide three times daily for at least 1 month followed by leuprolide or goserelin subcutaneously once monthly for four months. Beginning after the fourth administration of leuprolide or goserelin, patients undergo radiotherapy 5 days a week for 7-8 weeks. Beginning one month before radiotherapy and continuing until 1 month after radiotherapy, patients receive SU5416 IV over 60 minutes on days 1 and 4. Treatment repeats weekly in the absence of disease progression or unacceptable toxicity. Cohorts of 3-12 patients receive escalating doses of SU5416 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which at least 3 of 12 patients experience dose-limiting toxicity. Patients are followed every 4-6 weeks for 4 months and then every 8-12 weeks for 8 months.

PROJECTED ACCRUAL: A total of 3-18 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed adenocarcinoma of the prostate with at least 1 of the following: Clinical stage T2b or greater Gleason score at least 8 Pretreatment PSA greater than 15 ng/mL Pelvic and/or periaortic node(s) positive on abdominal/pelvic CT scan Metastatic disease requiring palliation for local symptoms No known brain metastases

PATIENT CHARACTERISTICS: Age: Not specified Performance status: ECOG 0-2 OR Karnofsky 60-100% Life expectancy: Not specified Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Platelet count at least 75,000/mm3 Hepatic: Bilirubin no greater than upper limit of normal (ULN) AST no greater than 2.5 times ULN Renal: Creatinine no greater than 1.5 mg/dL OR Creatinine clearance greater than 60 mL/min Cardiovascular: No symptomatic congestive heart failure No cardiac arrhythmia No uncompensated coronary artery disease on ECG or physical exam No myocardial infarction or severe unstable angina within the past 6 months No deep venous or arterial thrombosis within the past 3 months Pulmonary: No pulmonary embolism within the past 3 months Other: No other concurrent uncontrolled illness No ongoing or active infection No diabetes mellitus with severe peripheral vascular disease No psychiatric illness or social condition that would preclude study No prior allergic reactions attributed to compounds of similar chemical or biological composition to SU5416 or Cremophor EL vehicle No prior severe allergic reactions to paclitaxel or docetaxel

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: No concurrent anticancer chemotherapy Endocrine therapy: Prior hormonal therapy of any duration allowed Radiotherapy: No prior pelvic radiotherapy Surgery: No prior prostatectomy Other: No prior non-hormonal systemic therapy for prostate cancer No other concurrent investigational or commercial agents or therapies for malignancy No concurrent combination antiretroviral therapy for HIV-positive patients

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2001-11; Primary Completion 2002-03 (Actual); Study Completion 2003-04 (Actual)

PRIMARY OUTCOMES:
Side effects of SU5416 in combination with standard hormone treatment and radiation in men with prostate cancer | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Walter M. Stadler, MD, FACP, Study Chair — University of Chicago
Locations (3):
- United States (3):
  - Radiation Oncology, Chicago, Illinois
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - LaGrange Memorial Hospital, LaGrange, Illinois